CLINICAL TRIAL: NCT04818268
Title: Role of Sensory Working Memory in Speech Motor Learning Aim 2
Brief Title: Sensory Memory in Speech Motor Learning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: Yale University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025475_a; R01DC017439 (NIH)
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Speech; Consolidation
MeSH Terms: conditions — Speech | interventions — Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adaptation to Altered Auditory Feedback (Experimental): Adaptation to Altered Auditory Feedback
  Interventions: Behavioral: Adaptation
- Auditory Sensory Memory (Experimental): Auditory Sensory Memory
  Interventions: Behavioral: Adaptation
- Somatosensory Sensory Memory (Experimental): Somatosensory Sensory Memory
  Interventions: Behavioral: Adaptation
- Adaptation to Altered Auditory Feedback + cTBS to 46v (Experimental): Adaptation to Altered Auditory Feedback + cTBS to 46v
  Interventions: Behavioral: Adaptation; Other: cTBS
- Sensory Memory + cTBS to 46v (Experimental): Sensory Memory + cTBS to 46v
  Interventions: Behavioral: Adaptation; Other: cTBS

INTERVENTIONS:
Behavioral: Adaptation — Sensorimotor adaptation in speech
Other: cTBS — continuous theta-burst stimulation
  Arms: Adaptation to Altered Auditory Feedback + cTBS to 46v; Sensory Memory + cTBS to 46v

SUMMARY:
The proposed studies focus on memory for speech movements and sounds and its relation to learning. Continuous theta-burst transcranial magnetic stimulation (cTBS) will be used to suppress activity in a region of pre-frontal cortex associated with somatic and auditory working memory (Brodmann area 46v) to test its involvement in learning.

DETAILED DESCRIPTION:
This study will assess the relationship between sensory working memory and speech motor adaptation using a between subjects design. Participants will be assigned to one of two groups. Each group will undergo both auditory and somatosensory working memory tests. This will be followed by adaptation to altered auditory feedback. Using a different group of subjects, cTBS will be used to disrupt neural activity in Brodmann area 46v in ventrolateral prefrontal cortex to test its involvement in adaptation. One set of tests will focus on the effects of cTBS on both auditory and somatosensory working memory. A second set of tests will focus on the effects of cTBS on speech motor adaptation to altered auditory feedback. Both working memory and adaptation are assessed on 0 to 100 scales.

ELIGIBILITY:
Inclusion Criteria:

* right handed adults
* no known physical or neurological abnormalities

Exclusion Criteria:

* patients with:
* cardiac pacemaker
* surgical clips or values on the heart
* implants
* metal or metallic fragments in any part of the body
* pregnancy
* claustrophobia
* a personal or family history of epilepsy
* currently taking antipsychotic drugs
* currently taking antidepressant drugs
* currently taking antianxiety drugs
* history of concussion.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Speech Motor Learning | Performance as measured at the end of learning (single day experiment)
  Learning is assessed on a 0 to 100 scale as change in speech sounds (speech formant frequencies). A score of 100 corresponds to complete adaptation.
Sensory Memory | Single day experiment
  Sensory Memory is measured on a 0 to 100 scale. A score of 100 corresponds to perfect memory.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Haskins Laboratories
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04818268/ICF_000.pdf